CLINICAL TRIAL: NCT05595148
Title: Randomized Feasibility Trial for Immediate vs Delayed Weightbearing for Surgically Treated Fractures
Brief Title: Immediate Weightbearing vs Delayed Weightbearing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Robert O'Toole, Program Director, Orthopaedic traumatology, Director of Clinical Research, Department of Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00103274
Record Dates: First submitted 2022-10-10; First posted 2022-10-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Rehabilitation
Keywords: Feasibility; Orthopaedic trauma; randomized care; WBAT; Delayed weightbearing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate WBAT (Active Comparator): Recent studies have highlighted that early WBAT is may be safe following fixation of lower extremity, pelvis, and acetabulum fractures where the standard of care has been delayed WBAT, but high-quality prospective studies on this topic are needed.
  Interventions: Procedure: Immediate WBAT
- Delayed WBAT (Active Comparator): Though immediate postoperative WBAT has become the standard of care following fixation of pertrochanteric, femoral shaft, and tibial shaft fractures, most surgeons restrict patient weight bearing following fixation of other lower extremity and pelvis/acetabulum fractures. Progression to full weight bearing varies greatly by type of fracture, fixation method, and surgeon. Weight bearing restrictions following fracture fixation have been shown to be associated with various poor outcomes (increased complications, prolonged hospital length of stay, etc.), particularly in geriatric patients. Thus, it is important for us to understand if it is safe to allow early weight bearing following lower extremity and pelvis/acetabulum fracture fixation, as this could help expedite patient mobility and return to function, and potentially reduce complications.
  Interventions: Other: No Intervention: Delayed WBAT

INTERVENTIONS:
Procedure: Immediate WBAT — Men or women over 18 years who present with a fracture of the acetabulum, pelvis, distal femur, proximal tibia, distal tibia, who will undergo fracture fixation within 7 days of their injury and consent to the research study.
  Arms: Immediate WBAT
Other: No Intervention: Delayed WBAT — Patients with ankle fractures will be instructed to touch-down (toe touch or foot flat) weight bear (approximately 10% of body weight) while in the boot for. Patients will be instructed to keep foot off of floor or set ball of foot or heal on ground for balance using walker or crutches at all times. After the 6 week post op visit, patients may begin weight bearing as tolerated. Patients with tibial plateau fractures will be instructed to touch down (toe touch or foot flat) weight bear (approximately 10% of body weight) for at least 6 weeks. After the 6 week post op visit, patients may begin weight bearing as tolerated until full weight bearing is achieved.
  Arms: Delayed WBAT

SUMMARY:
The purpose of this study is to perform a feasibility trial of immediate versus delayed weight bearing following fixation of fractures of the lower extremity, pelvis, and acetabulum. The investigator will enroll patients from Shock Trauma over a period of 12 months, and randomize them to immediate weight bearing as tolerated (WBAT) versus delayed WBAT (non-weightbearing for 6-12 weeks). Four specific feasibility criteria will be assessed: enrollment (target 50%), follow-up (target 90% at 3 months), correct documentation of weight bearing (target 90%), correct documentation of primary outcomes, which include reoperation and hardware failure (target 90%). Target enrollment is patients with fractures where the current standard of care is delayed WBAT; for lower extremity this will include fractures of the distal femur, proximal tibia, and distal tibia, including select fractures with intra-articular extension. If feasibility criteria are met over the course of this study, the investigator hopes to move forward with a multicenter randomized controlled trial on this topic.

DETAILED DESCRIPTION:
Weight bearing restrictions are increasingly being scrutinized, as understanding of the potential negative effects of immobilization expand. Recent studies have highlighted that early WBAT may be safe following fixation of lower extremity, pelvis, and acetabulum fractures where the standard of care has been delayed WBAT, but high-quality prospective studies on this topic are needed.

The investigator hypothesizes that in a feasibility trial of immediate versus delayed WBAT following lower extremity, pelvis, and acetabulum fracture fixation, this trial will:

1. be able to enroll 50% of eligible patients and have a 90% follow-up at 90 days post-op of enrolled patients.
2. be able to achieve 90% correct documentation of postoperative weight bearing status and primary outcomes (reoperation or hardware failure).

Specific Aim 1 - Evaluate in a feasibility trial of immediate versus delayed WBAT following lower extremity, pelvis, and acetabulum fracture fixation whether 50% of patients can be enrolled, and 90% of those enrolled will have 90-day follow-up.

Specific Aim 2 - Evaluate in a feasibility trial of immediate versus delayed WBAT following lower extremity, pelvis, and acetabulum fracture fixation whether 90% correct documentation of postoperative weight bearing status and 90% correct documentation of primary outcomes (reoperation or hardware failure) can be obtained.

The investigator anticipates that the feasibility criteria will be met with regard to enrollment, follow-up, and documentation, which will allow us to begin a (likely multicenter) randomized controlled trial evaluating early versus delayed weight bearing following lower extremity, pelvis, and acetabulum fixation.

ELIGIBILITY:
Inclusion Criteria:

* Fracture of the acetabulum, pelvis, distal femur, distal tibia, including those with intra- articular extension, that meets surgical indications.
* Operative treatment within 7 days of injury at R Adams Cowley Shock Trauma Center, University of Maryland, University of Maryland Medical System, University of Maryland Capital Region Medical Center.
* Provision of informed consent.

Exclusion Criteria:

* Non English Speaking.
* Cognitive ability does not allow for full understanding of study procedures ( Patient has been diagnosed with psychiatric condition, intellectually challenged without adequate family support).
* Patient has other orthopaedic or non-orthopaedic injuries that would preclude him/her from being able to weight bear immediately (e.g. open fractures, polytrauma.
* Significant impaction (>2mm) or comminution at joint surface (e.g. with acetabulum, distal femur, tibial plateau, or tibial plafond fractures).
* Patients who would not be able to immediately weight bear or comply with weight bearing restrictions.
* Not willing to be randomized.
* Surgeon or clinical follow will not occur at participating hospital or location.
* Anticipated problems with follow up in the judgement of study personnel ( patient is homeless).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The number of participants with unplanned reoperation or hardware failure | 6 months following definitive fixation surgery
  Any reoperation associated with the enrolled fracture region (non union, malunion, hardware removal)

SECONDARY OUTCOMES:
Percentage of patients who maintained follow-up | 12 months following definitive fixation surgery
  Greater than 80% of enrolled patients maintained followup for 12 months following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Robert O'Toole, MD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland, Shock Trauma Center, Baltimore, Maryland
  - University of Maryland, Capital Region Health, Cheverly, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunningham BP, Ali A, Parikh HR, Heare A, Blaschke B, Zaman S, Montalvo R, Reahl B, Rotuno G, Kark J, Bender M, Miller B, Basmajian H, McLemore R, Shearer DW, Obremskey W, Sagi C, O'Toole RV. Immediate weight bearing as tolerated (WBAT) correlates with a decreased length of stay post intramedullary fixation for subtrochanteric fractures: a multicenter retrospective cohort study. Eur J Orthop Surg Traumatol. 2021 Feb;31(2):235-243. doi: 10.1007/s00590-020-02759-3. Epub 2020 Aug 14. PMID 32797351
- [Background] Gaski GE, Manson TT, Castillo RC, Slobogean GP, O'Toole RV. Nonoperative treatment of intermediate severity lateral compression type 1 pelvic ring injuries with minimally displaced complete sacral fracture. J Orthop Trauma. 2014 Dec;28(12):674-80. doi: 10.1097/BOT.0000000000000130. PMID 24740110
- [Background] Gitajn IL, Connelly D, Mascarenhas D, Breazeale S, Berger P, Schoonover C, Martin B, O'Toole RV, Pensy R, Sciadini M. Is prescribed lower extremity weight-bearing status after geriatric lower extremity trauma associated with increased mortality? Injury. 2018 Feb;49(2):404-408. doi: 10.1016/j.injury.2017.12.012. Epub 2017 Dec 14. PMID 29249533
- [Background] Marchand LS, Horton S, Mullike A, Goel R, Krum N, Ochenjele G, O'Hara N, O'Toole RV, Eglseder WA, Pensy R. Immediate Weight Bearing of Plated Both-Bone Forearm Fractures Using Eight Cortices Proximal and Distal to the Fracture in the Polytrauma Patient Is Safe. J Am Acad Orthop Surg. 2021 Aug 1;29(15):666-672. doi: 10.5435/JAAOS-D-20-01252. PMID 34030171
- [Derived] Mittwede PN, Li V, Okhuereigbe DO, Bell AC, Loudermilk C, Demyanovich HK, Lawrence JE, Turner KE, Kovvur M, Brand JP, Cunningham DJ, Johnson DJ, Sepehri A, Sciadini MF, Nascone JW, Gage MJ, Hempen EC, O'Hara NN, Slobogean GP, O'Toole RV. Immediate versus delayed weight bearing for fractures of the pelvis, acetabulum, distal femur, and proximal and distal tibia: a feasibility randomized controlled trial. Pilot Feasibility Stud. 2025 Nov 5;11(1):133. doi: 10.1186/s40814-025-01708-3. PMID 41194216